CLINICAL TRIAL: NCT05756127
Title: Predicting Incident Heart Failure from Population-based Nationwide Electronic Health Records: Protocol for a Model Development and Validation Study
Brief Title: Future Innovations in Novel Detection of Heart Failure FIND-HF
Acronym: FIND-HF
Status: Active, not recruiting | Type: Observational
Sponsor: University of Leeds (Other)
Collaborators: Japan Foundation for Aging and Health (Other)
Responsible Party: Principal Investigator, Dr Christopher Gale, Professor of Cardiovascular Medicine, University of Leeds
Other Study IDs: FINDHF01
Record Dates: First submitted 2023-01-31; First posted 2023-03-06 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure
Keywords: heart failure; Prediction model
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All eligible patients: Observational cohort using anonymized patient-level primary care data linked to secondary administrative data; CPRD-GOLD and CPRD-AURUM.
  Interventions: Other: Observational - no intervention given

INTERVENTIONS:
Other: Observational - no intervention given — Observational - no intervention given

SUMMARY:
Heart failure (HF) is increasingly common and associated with excess morbidity, mortality and healthcare costs. New medications are now available which can alter the disease trajectory and reduce clinical events. However, many cases of HF remain undetected until presentation with more advanced symptoms, often requiring hospitalisation. Earlier identification and treatment of HF could reduce downstream healthcare impact, but predicting HF incidence is challenging due to the complexity and varying course of HF. The investigators will use routinely collected hospital-linked primary care data and focus on the use of artificial intelligence methods to develop and validate a prediction model for incident HF. Using clinical factors readily accessible in primary care, the investigators will provide a method for the identification of individuals in the community who are at risk of HF, as well as when incident HF will occur in those at risk, thus accelerating research assessing technologies for the improvement of risk prediction, and the targeting of high-risk individuals for preventive measures and screening.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 16 years and older
2. No history of heart failure
3. A minimum of one year follow up

Exclusion Criteria:

-

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will comprise all available patients in CPRD-GOLD who were eligible for data linkage and had at least 1-year follow-up in the period between 2nd Jan 1998 and 28th February 2022. The outcome of interest is the first diagnosed HF, and will be identified using Read codes (for the CPRD patient profile) and ICD-10 codes (for HES events). Patients with less than one year of registration in CPRD, those who are under eighteen years of age at the date of the first registration in CPRD, those who were diagnosed with HF before 2nd Jan 1998, and those who were not eligible for data linkage will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 14000 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To develop and validate a for predicting the risk of new onset HF | Between 2nd Jan 1998 and 28 Feb 2022
  Predictive factors will be identified using Read codes (diagnoses), All variables will be considered as potential predictors, and may include:
  1. sociodemographic variables: age, sex, ethnicity, index of multiple deprivation;
  2. lifestyle factors (e.g. smoking status, alcohol consumption);
To identify and quantify the magnitude of predictors of new onset HF | Between 2nd Jan 1998 and 28 Feb 2022
  The proposed model can extract informative risk factors from EHR data. Specifically we will fit multivariable Cox proportional hazard models with backwards elimination approach to retain predictors of incident HF within each prediction window.

CONTACTS AND LOCATIONS:
Overall Officials: Chris P Gale, Principal Investigator — University of Leeds
Locations (1):
- University of Leeds, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nakao YM, Nadarajah R, Shuweihdi F, Nakao K, Fuat A, Moore J, Bates C, Wu J, Gale C. Predicting incident heart failure from population-based nationwide electronic health records: protocol for a model development and validation study. BMJ Open. 2024 Jan 22;14(1):e073455. doi: 10.1136/bmjopen-2023-073455. PMID 38253453